CLINICAL TRIAL: NCT04632082
Title: A Pragmatic Superiority Randomized Controlled Trial Comparing Telepsychoeducation Plus Personalized Videos vs. Telepsychoeducation Without Personalized Videos for the Prevention of Future Emotional Distress in Professionals From Essential Services With Low to Moderate Levels of Emotional Distress in Brazil in the Context of COVID-19
Brief Title: Telepsychoeducation for the Prevention of Emotional Distress in Professionals and Students From Essential Services in the Context of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Giovanni Abrahao Salum Junior, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20200213_Prevention
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Mental Health Wellness 1; COVID; Emotional Distress; Depressive Symptoms; Anxiety Symptoms; Irritability; Telepsychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two-group randomized clinical trial including health professionals and health students suffering from low to moderate levels of anxiety, depression and irritability symptoms during the COVID-19 outbreak, randomized randomized 1:1 to the Telepsychoeducation with personalized videos (2 sessions with a psychologist plus 2 videos a week for 4 weeks chosen based on symptom presentation) or Telepsychoeducation without personalized videos (2 sessions with a psychologist focused on reassurane and aspects of the outbreak).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Telepsychoeducation with personalized videos (Experimental): One psychoeducation session administered by a therapist by video call, with interventions focused on promoting protective factors and reducing common risk factors for psychopathology. The intervention is complemented by the sending of 4 videos of 2 to 3 minutes, with psychoeducational content, sent each week by the therapist.
  Interventions: Behavioral: Telepsychoeducation with personalized videos
- Comparator: Telepsychoeducation without personalized videos (Active Comparator): One psychoeducation session administered by a therapist by video call, with interventions focused on promoting protective factors and reducing common risk factors for psychopathology.
  Interventions: Behavioral: Telepsychoeducation without personalized videos

INTERVENTIONS:
Behavioral: Telepsychoeducation with personalized videos — 1 session with a psychologist plus 1 video a week for 4 weeks chosen based on symptom presentation
  Arms: Intervention: Telepsychoeducation with personalized videos
Behavioral: Telepsychoeducation without personalized videos — 1 session with a psychologist focused on reassurance and aspects of the outbreak
  Arms: Comparator: Telepsychoeducation without personalized videos

SUMMARY:
A pragmatic superiority randomized controlled trial comparing Telepsychoeducation plus personalized videos vs. Telepsychoeducation without personalized videos for the prevention of future emotional distress in professionals and students from essential services with low to moderate levels of emotional distress in Brazil.

Note: This study was approved by the Ethics and Research Committee of the Hospital de Clínicas de Porto Alegre and is originally registered at Plataforma Brasil, a Brazilian study registration platform (under CAAE: 30608420.5.0000.5327). Recruitment began in May 28th 2020.

DETAILED DESCRIPTION:
TITLE: "A pragmatic superiority randomized controlled trial comparing Telepsychoeducation plus personalized videos vs. Telepsychoeducation without personalized videos for the prevention of future emotional distress in professionals and students from essential services with low to moderate levels of emotional distress in Brazil"

IMPORTANCE: COVID-19 outbreak is associated with increased emotional distress (depression, anxiety and irritability) all over the world. Currently, there are no large randomized trials testing preventive interventions to reduce the burden caused by mental disorders after the occurrence of a pandemic outbreak in these proportions.

OBJECTIVE: To compare the effectiveness of Telepsychoeducation with personalized videos to Telepsychoeducaton without personalized videos for the prevention of severe symptoms of emotional distress (anxiety, depression and irritability) in health professionals with a low to moderate level of those symptoms in Brazil during the COVID-19 outbreak.

DESIGN, SETTING, AND PARTICIPANTS Two-group randomized clinical trial. Participants were recruited in Brazil from the national service of telehealth provided by the ministry of health. Participants included health professionals suffering from low to moderate levels of anxiety, depression and irritability symptoms during the COVID-19 outbreak. Low to moderate levels of symptoms were defined by all of the following: (1) z score lower than 1.5 on the PROMIS Anxiety Scale; (2) z score lower than 1.5 on the PROMIS Depression Scale; (3) z score lower than 1.5 on the PROMIS Anger Scale.

INTERVENTIONS: All participants were randomized to the Telepsychoeducation with personalized videos (1 session with a psychologist plus 1 videos a week for 4 weeks, chosen based on symptom presentation) or Telepsychoeducation without personalized videos (1 session with a psychologist focused on reassurance and aspects of the outbreak).

MAIN OUTCOMES AND MEASURES: The primary outcome will be the proportion of participants with a T score equal or above 70 in any of the emotional distress scales (anxiety, depression or irritability) in 6 months. Secondary outcomes (1) mean score change in individual scales at 1, 3 and 6 months; (2) proportion of participants with a T score equal or above 60 in any of the emotional distress scales at 1, 3 and 6 months; and (3) service satisfaction and net-promoter score at the end of the treatment.

EXPECTED RESULTS: To detect a 5% group difference between each group, an alpha of 0.05, power of 90% and 20% loss to follow up, in a 1:1 randomization, we would need a total of 1100 participants per group.

ELIGIBILITY:
Inclusion Criteria (must present all of the following):

Professionals and students from essential services suffering from low to moderate emotional distress

* z score lower than 1.5 on the PROMIS Anxiety Scale
* z score lower than 1.5 on the PROMIS Depression Scale
* z score lower than 1.5 on the PROMIS Anger Scale

Exclusion Criteria:

* Moderate to severe suicide risk assessed by a psychiatrist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-07-13 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
Incident Cases in 6 months | 6-months
  Proportion of participants with a T score equal or above 70 in any of three emotional distress subscales (Patient-Reported Outcomes Measurement Information System - or PROMIS - of Depression, Anxiety and Anger)

SECONDARY OUTCOMES:
Incident cases | 1, 3 an 6-months
  Proportion of participants with a T score equal or above 60 in any of the emotional distress scales (PROMIS - of Depression, Anxiety and Anger)
Service Satisfaction | 2-weeks
  Service satisfaction measured by the net-promoter score at the end of the treatment (proportion of promoters - scores of 9 or 10)
Improvement in Quality of Life | 1, 3 and 6-months
  Mean score change in quality of life scale (PROMIS General Life Satisfaction Scale or GLSS)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Salum, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre, Porto Alegre/Brazil
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to share study protocol, SAP, ICF, CRS, analytic code and individual-based variables.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Avaliable six months after study completion (antecipated - January 2022)
Access Criteria: Researchers and civil society

REFERENCES:
- [Derived] Damiano RF, Abreu M, Dreher CB, Bryan CJ, Miguel EC, Fleck M, Manfro GG, Salum GA. Risk Factors for Suicide Attempts and Psychiatric Hospitalization Among Brazilian Health Care Professionals. J Clin Psychiatry. 2025 Dec 31;87(1):25m15858. doi: 10.4088/JCP.25m15858. PMID 41499179
- [Derived] Salum GA, Spanemberg L, Costa MA, Simioni AR, Gosmann NP, Hartmann de Souza L, Cuijpers P, Pine DS, Brunoni AR, Katz N, Umpierre RN, Kristensen CH, Manfro GG, Fleck MP, Dreher CB. Single-session intervention with and without video support to prevent the worsening of emotional distress among healthcare workers during the SARS-CoV-2 pandemic: a randomised clinical trial. BMJ Ment Health. 2025 Apr 7;28(1):e301416. doi: 10.1136/bmjment-2024-301416. PMID 40194849
- [Derived] Costa MA, Kristensen CH, Dreher CB, Manfro GG, Salum GA. Habituating to pandemic anxiety: Temporal trends of COVID-19 anxiety over sixteen months of COVID-19. J Affect Disord. 2022 Sep 15;313:32-35. doi: 10.1016/j.jad.2022.06.077. Epub 2022 Jun 27. PMID 35772625